CLINICAL TRIAL: NCT02884362
Title: Creation of a Prospective Melanoma Database
Brief Title: Prospective Melanoma Database
Status: Recruiting | Type: Observational
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Other Study IDs: 16HLCUTA01
Record Dates: First submitted 2016-07-28; First posted 2016-08-31 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-07

CONDITIONS: Melanoma
Keywords: melanoma clinical biological database
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor sample
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: clinical biological data collection on melanoma — collection and centralization of clinical and biological data of patients with melanoma

SUMMARY:
In research on melanoma, translational research is the essential link between basic research and clinical research by facilitating the passage between discovery and improvement in the quality of patients care.That is the reason why it is very important to collect, and centralize clinical and biological data of patients with melanoma.

The aim of the project is to provide to scientific community a structured, mixed clinical and biological database, unique in France, in order to insure accessibility to clinical data.

DETAILED DESCRIPTION:
collection of clinical and biological data from patients with melanomas of any stage in a structured and centralized database

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Histologically confirmed melanoma of any stage
* Affiliated to a social security system in france
* Who signed the informed consent

Exclusion Criteria:

* Any psychiatric or medical condition that would make the patient unable to give a signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with any histological type of melanoma and of any stage
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2016-01; Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Database of patients with melanoma | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MEYER, MD PHD, Principal Investigator — Institut claudius regaud Toulouse ONCOPOLE
Locations (1):
- Institut claudius regaud IUCT ONCOPOLE, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided